CLINICAL TRIAL: NCT02197650
Title: Expanded Access Program for a Multicentre, Open, Non Randomized Study, Evaluating Safety of Erythrocytes Encapsulating L-asparaginase (GRASPA®) in Combination With Polychemotherapy in Patients Under 55 Years Old With Acute Lymphoblastic Leukemia (ALL) at Risk to Receive Other Formulation of Asparaginase
Brief Title: Expanded Access Program: Safety of Erythrocytes Encapsulating L-asparaginase (GRASPA®) in Combination With Polychemotherapy in Patients Under 55 Years Old With Acute Lymphoblastic Leukemia (ALL) at Risk to Receive Other Formulation of Asparaginase
Acronym: EAP
Status: No longer available | Type: Expanded Access
Sponsor: ERYtech Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: GRASPALL 2012-10-EAP
Record Dates: First submitted 2014-05-07; First posted 2014-07-23 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL L-asparaginase encapsulated erythrocytes
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — eryaspase

INTERVENTIONS:
Drug: suspension of erythrocytes encapsulating L-asparaginase — Erythrocytes encapsulating L-asparaginase
  Other Names: GRASPA®; eryaspase

SUMMARY:
Early Access Program to provide L-asparaginase encapsulated in Erythrocyte (GRASPA®) for patient unable to receive any other form of Asparaginase.

DETAILED DESCRIPTION:
Some patients can not be eligible to other clinical trials / program sponsored by Erytech Pharma but could have a benefit to be treated with GRASPA. Following discussion with French regulatory authorities, it has been suggested to propose access to GRASPA to patients unable to receive any other form of L-asparaginase and not eligible to the ongoing study or other program. This exploratory study should allow it in an "Expended Access Program" framework.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ALL de novo or in relapse or refractory
* Eligible to a chemotherapy treatment including L-asparaginase
* Known contraindication and/or at risk of toxicity to other L-asparaginase formulation according to investigator opinion based on information available
* Patient under 55 years old
* Patient informed and consent provided (the 2 parents need to consent for children).

Exclusion Criteria:

* Patient unable to receive GRASPA due to general or visceral conditions

  * Serum creatinine ≥ 2 x ULN unless related to ALL
  * ALT or AST ≥ 3 x ULN unless related to ALL
  * Active clinical pancreatitis any grade or pancreatic enzyme elevation ≥ 1.5 ULN
  * Other serious conditions according to investigator's opinion.
* Absence of documented serological test for HIV, B and C hepatitis
* History of grade 3 transfusional incident or any contraindication to receive blood transfusion
* Patient under concomitant treatment likely to cause hemolysis
* Presence of specific anti-erythrocyte antibodies preventing from getting a compatible erythrocyte concentrate for the patient.
* Patient undergoing yellow fever vaccination.
* Patient under phenytoin treatment.
* Women of childbearing potential without effective contraception as well as pregnant or breast feeding women.
* Patient already included in another clinical trial

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pr. Yves BERTRAND, Principal Investigator — IHOP, Lyon; Pr. Hervé DOMBRET, Principal Investigator — Hôpital Saint Louis Paris
Locations (10):
- France (10):
  - Hôpital Jean Minjoz - Batiment MEMCP, Besançon
  - CHRU Lille - Hôpital Claude-Huriez, Lille
  - IHOP, Lyon
  - Hôpital de l'Archet 2, Nice
  - Hôpital Saint Louis, Paris
  - CHU Rouen - Hôpital des enfants, Rouen
  - CHU Saint Etienne Hôpital Nord, Saint-Etienne
  - Institut Universitaire du Cancer, Toulouse
  - Hôpital BRETONNEAU, Tours
  - Hôpital Brabois Enfants, Vandœuvre-lès-Nancy